CLINICAL TRIAL: NCT06325670
Title: Better Treatment of Patients With Type 2 Diabetes and Binge Eating Disorder (BED)
Brief Title: Type 2 Diabetes and Binge Eating Disorder (BED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Jascha Fonden (Other); Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23/50374
Record Dates: First submitted 2024-03-01; First posted 2024-03-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Binge-Eating Disorder
Keywords: BED; T2D; Treatment; Binge Eating Disorder; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Binge-Eating Disorder; Diabetes Mellitus | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BED treatment (Experimental): The BED group therapy program consists of 11 sessions, followed by a 3-month follow-up session. Each 3-hour session accommodates eight patients and two psychologists. Treatment follows a manualized cognitive behavioral therapy approach, with patients receiving a complimentary manual at the start. Sessions are conducted both in-person and online using a blended care model, with about one-third delivered virtually.
  Interventions: Behavioral: BED treatment
- Waitlist (Other): The waitlist control group consists of participants who are placed on a waiting list to receive treatment. While participants in the treatment group immediately receive BED treatment (Arm 1), those in the waitlist control group do not receive active treatment initially. They remain on the waiting list for 6 months until the treatment group completes their intervention. At that point, participants in the waitlist control group also receive the same BED treatment, serving as a comparison group to evaluate the intervention's effectiveness.
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: BED treatment — A 12 session cognitive behavioural intervention in groups for Danish adults with type 2 diabetes and Binge Eating Disorder.
  Arms: BED treatment
Other: Waitlist — A waitlist control group that receives regular type 2 diabetes treatment while waiting to receive the BED treatment intervention.
  Arms: Waitlist

SUMMARY:
The goal of this research project is to improve the treatment of individuals living with both type 2 diabetes (T2D) and Binge Eating Disorder (BED). The research hypothesizes that BED treatment will not only improve BED symptoms but also improve T2D severity and associated cardiovascular risk factors. The research involves a multidisciplinary team, including experts in endocrinology, psychology, and eating disorders.

The main questions it aims to answer are:

* Does treatment for Binge Eating Disorder lead to improvements in BED symptoms?
* Does treatment for Binge Eating Disorder lead to improvements in T2D severity and associated cardiovascular risk factors?

Participants will undergo a comprehensive treatment program targeting both BED and T2D. This program will include psychotherapy sessions focusing on cognitive-behavioral techniques to address binge eating behavior.

Researchers will compare participants' outcomes before and after the treatment program to assess changes in BED symptoms, T2D severity, and associated cardiovascular risk factors.

DETAILED DESCRIPTION:
This research project aims to address the treatment challenges faced by individuals living with both type 2 diabetes (T2D) and Binge Eating Disorder (BED). It is estimated that approximately 300,000 people in Denmark have T2D, while 40-50,000 adults suffer from BED. The prevalence of BED among patients with T2D is up to 20%, and individuals with T2D and BED often experience more somatic and psychological symptoms compared to those with T2D alone.

The primary objective of this project is to improve the treatment outcomes for patients with coexisting T2D and BED. To achieve this, the project has three specific aims:

1. Prevalence assessment: The project aims to identify the prevalence of BED within a cohort of approximately 4,000 patients diagnosed with T2D in the Region of Southern Denmark. This cohort is part of the DD2 cohort, managed by the Danish Center for Strategic Research in Type 2 Diabetes.
2. Treatment efficacy investigation: The project will conduct a Randomized Controlled Trial (RCT) involving 64 patients diagnosed with both T2D and BED. The trial will investigate the effects of BED treatment on various outcomes, including changes in BED symptoms, glycemic control, and associated cardiovascular risk factors.
3. Glucose sensor study: Patients will be assessed using continuous glucose monitoring sensors for a week before and after pre- and post-test visits at Odense University Hospital (OUH). This allows for detailed blood glucose profiles without finger pricking. Data on time in range, time below range, variability, and area under the curve will be extracted from the sensors. These data aim to provide insights into glycemic variability, complementing traditional HbA1c measurements and aiding in evaluating the intervention's effectiveness.

By addressing these aims, the project seeks to enhance the understanding of the prevalence of BED among individuals with T2D and evaluate the efficacy of BED treatment interventions in improving health outcomes for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* A diagnosis of mild to severe BED based on thorough assessment
* Sufficient ability to communicate in Danish
* Ability to sit on a chair for up to 3 hours

Exclusion Criteria:

* Previously diagnosed with autism spectrum disorder or psychotic disorders
* Dementia or developmental disability.
* Severe anxiety or depression or personality disorder assessed through clinical interview with SCID (based on DSM-V criteria)
* Currently experiencing severe to moderate substance abuse

Use of weight loss medication is not an exclusion criterion but is clearly noted regarding the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2026-02-03 (Actual)

PRIMARY OUTCOMES:
Number of binge eating episodes | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks after for 7 days), and follow up (three months)
  This outcome will assess changes in the number of binge eating episodes per week among participants receiving BED treatment compared to baseline

SECONDARY OUTCOMES:
Binge Eating Disorder Questionnaire | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks), and follow up (three months)
  BED-Q is a questionnaire consisting of 10 items, with questions 1-7 assessed on a Likert scale from 0-5. Together, these questions constitute a score ranging from 0-35, indicating the severity of Binge Eating Disorder (BED) from none to mild, moderate, severe, and extreme. The items in BED-Q are carefully crafted to reflect the diagnostic criteria for Binge Eating Disorder (BED) according to DSM-5, including (1) episodes of binge eating large amounts of food in a short period (within two hours); (2) a sense of losing control over eating; (3) eating faster than usual; (4) eating until uncomfortably full; (5) eating when not hungry; (6) eating alone; and (7) experiencing negative emotions such as guilt or shame after binge eating. Question 8 is used to screen for any compensatory behaviors, such as vomiting, while questions 9 and 10 examine the distress associated with binge eating episodes.
Glucose Sensor Data for Blood Glucose Profile | Baseline (Days 0-7), post treatment/post waitlist (up to 20 weeks after for 7 days)
  Glucose sensor data will be collected using continuous glucose monitoring devices to assess blood glucose profiles during the first week and the last week of the treatment period. This non-invasive method captures real-time glucose levels over time, providing insights into glucose variability and trends. The collected data will aid in evaluating the effectiveness of the intervention in managing blood glucose levels and overall glycemic control.
HbA1c | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks)
  HbA1c, or glycated hemoglobin, levels are measured as a blood sample (2 ml) to assess long-term blood sugar control. This measure reflects average blood glucose levels over the past two to three months, and lower HbA1c levels indicate better glycemic control.

OTHER OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks)
  EDE-Q is a self-report questionnaire used to assess symptoms of eating disorders, particularly anorexia nervosa, bulimia nervosa, and Binge Eating Disorder (BED). It comprises various questions covering areas such as eating disorder symptoms, eating behaviors, and thoughts about body and weight. Participants complete the questionnaire to provide information about their eating patterns and body image.
Major Depression Inventory (MDI) | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks)
  The Major Depression Inventory (MDI) is a self-report questionnaire designed to assess the presence and severity of symptoms of major depression. It consists of 10 questions covering various aspects of depression, such as mood, energy level, concentration, sleep patterns, and appetite changes. Participants respond to the questions using a 6-point Likert scale ranging from 0 to 5. The total score ranges from 0 to 50, with a higher score reflecting more symptoms of depression.
Problem Areas In Diabetes (PAID20) | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks)
  PAID20 is a validated and extensively tested 20-item questionnaire that quantifies the emotional burden experienced by individuals with diabetes. This includes feelings of guilt, frustration, worry, and self-blame related to their diabetes. PAID questions are measured on a 5-point Likert scale with response options ranging from 0 to 4. PAID20 has demonstrated sensitivity to changes over time, making it suitable for evaluating the impact of therapeutic interventions and treatments in individuals with diabetes.
Lipid profile | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks)
  Lipid profile assessments is measured as a blood sample (3 ml) and includes various blood lipid levels; cholesterol, triglycerides, and lipoproteins. Cholesterol levels, including HDL (high-density lipoprotein) and LDL (low-density lipoprotein), are evaluated to assess lipid metabolism and cardiovascular risk.
Body Mass Index (BMI) | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks)
  BMI will be calculated as an outcome measure by combining weight (measured in kilograms) and height (measured in centimeters). BMI is calculated by dividing weight by the square of height. Participants are provided with blinded weighings, as weight loss is not the target of our intervention.
Blood Pressure | Baseline (Day 0), post treatment/post waitlist (up to 20 weeks)
  Blood pressure assessments will be conducted to evaluate cardiovascular health. Measurements will include systolic and diastolic pressures, recorded in millimeters of mercury (mmHg), to assess overall cardiovascular function and risk of cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Fiil Nybo, cand.psych., Principal Investigator — University og Southern Denmark, SDU; Jakob Linnet, Dr.med., cand.psych., Principal Investigator — Occupational- and Environmental Clinic, OUH; Michael Roeder, Dr.med., Principal Investigator — Steno Diabetes Center Odense
Locations (1):
- Region Of Southern Denmark Locations, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT06325670/SAP_000.pdf